CLINICAL TRIAL: NCT00009763
Title: Combined Modality Radioimmunotherapy For Metastatic Breast Adenocarcinoma With Two Cycles Of Escalating Dose 90Y-DOTA-peptide-m170 and Fixed, Low Dose Paclitaxel With Blood Stem Cell Support And Cyclosporin For HAMA Suppression
Brief Title: Monoclonal Antibody Therapy, Cyclosporine, and Paclitaxel in Treating Patients With Recurrent or Refractory Metastatic Breast Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, Davis (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068369; UCD-992080; NCI-V00-1640
Record Dates: First submitted 2001-02-02; First posted 2003-01-27 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2003-11

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Filgrastim; M1-70 monoclonal antibody; Cyclosporine; Paclitaxel; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Biological: monoclonal antibody m170
Drug: cyclosporine
Drug: paclitaxel
Procedure: peripheral blood stem cell transplantation
Radiation: yttrium Y 90 monoclonal antibody m170

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining monoclonal antibody therapy with cyclosporine and paclitaxel may be an effective treatment for metastatic breast cancer.

PURPOSE: Phase I trial to study the effectiveness of radiolabeled monoclonal antibody therapy, cyclosporine, and paclitaxel in treating patients who have recurrent or refractory metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of yttrium Y 90 monoclonal antibody m170 in combination with cyclosporine and paclitaxel in patients with recurrent or refractory metastatic breast cancer.
* Determine the preliminary efficacy of this regimen in these patients.

OUTLINE: This is a dose-escalation study of yttrium Y 90 monoclonal antibody m170 (Y90 MOAB m170).

Patients receive filgrastim (G-CSF) subcutaneously (SC) daily for 4 days prior to apheresis which continues daily for a maximum of 5 days. A minimum of 6 million CD34+ cells/kg must be harvested.

Patients receive oral cyclosporine every 12 hours on days -3 to 25. Patients receive unlabeled monoclonal antibody (MOAB) m170 IV followed by a tracer dose of indium In 111 MOAB m170 IV on day 0. On day 7, patients receive unlabeled MOAB m170 IV followed by Y90 MOAB m170 IV. Patients in cohorts 2-4 also receive paclitaxel IV over 3 hours on day 9.

If needed, patients undergo autologous peripheral blood stem cell transplantation on day 21 and receive G-CSF SC daily until blood counts recover.

Cohorts of 3-6 patients receive escalating doses of Y90 MOAB m170 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed monthly for 3 months, every 3 months for 1 year, and then every 6 months for 1 year.

PROJECTED ACCRUAL: A total of 18-30 patients will be accrued for this study within 36 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic breast adenocarcinoma

  * Residual or recurrent disease after first-line standard chemotherapy
  * Clinical evidence of metastatic disease
* Tumor cells positive for m170 immunoreactivity
* HAMA titer negative
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Not specified

Menopausal status:

* Not specified

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL

Renal:

* Creatinine less than 1.5 mg/dL

Cardiovascular:

* LVEF at least 50% by MUGA

Pulmonary:

* FEV1 at least 65% of predicted
* FVC at least 65% of predicted
* DLCO at least 60%

Other:

* No other malignancy within the past 5 years except nonmelanoma skin cancer or adequately treated carcinoma in situ of the cervix
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Chemotherapy

Chemotherapy:

* See Disease Characteristics
* At least 1 prior chemotherapy regimen for advanced disease
* Prior high-dose chemotherapy with autologous stem cell transplantation is allowed if given at least 12 months prior to study and carmustine was not used
* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior external beam radiotherapy
* No prior radiotherapy to more than 25% of the total skeleton

Surgery:

* Not specified

Other:

* No requirement for oral anticoagulants (low-dose warfarin for central line thrombosis prophylaxis allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-03

CONTACTS AND LOCATIONS:
Overall Officials: Carol M. Richman, MD, Study Chair — University of California, Davis
Locations (1):
- University of California Davis Cancer Center, Sacramento, California, United States